CLINICAL TRIAL: NCT04629742
Title: A Lower Sodium Neapolitan Pizza Prepared With Seawater in Place of Salt: Nutritional Properties, Sensory Characteristics and Metabolic Effects
Brief Title: Low Sodium Neapolitan Pizza Prepared With Seawater: Nutritional Properties, Sensory Characteristics, Metabolic Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Strazzullo, Principal investigator, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 403.20
Record Dates: First submitted 2020-10-29; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Satiety Response; Carbohydrate Metabolism; Sodium Retention
Keywords: salt reduction; seawater; pizza; hedonic food; water and sodium handling
MeSH Terms: conditions — Hypernatremia

STUDY DESIGN:
Intervention Model Description: Twelve healthy volunteers were recruited for a Randomized Controlled Trial, with the consumption of one Standard Pizza and one seawater pizza using a balanced crossover design, with 1 week wash out
Who Masked: Participant, Care Provider, Investigator
Masking Description: Nobody (unless the principal investigator) knows the types of pizza and their coding system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seawater Pizza (Experimental): Administration of a seawater pizza
  Interventions: Other: Seawater Pizza
- Standard Pizza (Active Comparator): Administration of a Standard pizza
  Interventions: Other: Standard pizza

INTERVENTIONS:
Other: Seawater Pizza — A seawater pizza administered to 12 healthy subjects
  Arms: Seawater Pizza
Other: Standard pizza — A standard pizza administered to 12 healthy subjects
  Arms: Standard Pizza

SUMMARY:
Seawater is rich in minerals which may help confer good palatability to foods, favouring the use of smaller amounts of salt, a recognized measure of cardiovascular prevention. The aim of this study is to investigate the nutritional properties, sensory characteristics and metabolic effects of a typical Neapolitan pizza prepared with seawater (SWP) in place of common salt, in comparison with Standard traditional Pizza (StP). Methods: The nutritional characteristics and the chemical profile of the SWP and StP were assessed by chemical analyses and the use of Food Composition Tables. Twelve healthy volunteers will be recruited for a Randomized Controlled Trial, with the consumption of one StP and one SWP using a balanced crossover design. The satiating power and palatability of the two pizzas will be tested by the administration of Visual Analogue Scales. Serum glucose, insulin and sodium will be measured every 30 minutes and 3-hour urines will be collected after each meal.

DETAILED DESCRIPTION:
The aim of the present study is testing the nutritional properties, the sensory characteristics and the metabolic effects of a novel recipe of Neapolitan pizza featuring the substitution of common salt with commercial seawater in such proportion as to reduce the total amount of sodium chloride in the otherwise traditional dough by approximately 50%.

The dough for both StP and SWP will be prepared from 170 g of organic flour (Agguggiaro and Figna 5 stagioni, 80% type 00/20% type 1, Curatolo, Padova, Italy) with the addition of 110 mL of tap water or commercial seawater respectively. To the StP 0.05 g of brewer's yeast and 5 g of unrefined salt (Sale Vero, Oro di Sicilia Srl, Nubia di Paceno, Trapani, Italy) will be added, while only 0.02 g of yeast and no salt were added to the SWP. Because salt is known to reduce the fermentation rate, based on the calculation that the amount of sodium chloride in SWP would be approximately one half of the StP content, it was decided to use approximately half the amount of yeast while maintaining constant the fermentation time, which was 15 h for both doughs. Commercial seawater is supplied by Steralmar Srl (Bisceglie, BT, Italia).

The trial is conceived as a double blind balanced randomised crossover trial, where each subject acted as his/her own control by consuming the two different pizzas at one week elapsed time from one another according to a balanced randomised sequence. The trial was approved by the Ethical Committee of the University of Naples Federico II (n. 403.20).

The participants will sign an informed consent to participate and receive detailed written instructions by a trained researcher about the study protocol: avoid any intense physical activity and complete the evening meal by 9 pm on the day before the test; have a standard breakfast (explained in detail) before 8.30 on the morning of the test; drink at least 300 mL of water between breakfast and the meal test, to guarantee normal hydration, not eating between breakfast and the meal test to guarantee a standard hunger level.

Weight, height and blood pressure (BP) will be measured just before the test, systolic and diastolic blood pressure and heart rate will be measured 3 times and the participants will be requested to void just before being weighted and the urines produced thereafter during the 3 h of the test will be collected.

The meals will be consumed in groups of 4 volunteers at a time under standard conditions in the metabolic kitchen at Federico II University Hospital.

The volunteers will be requested to drink 300 mL of water during the meal, which will have a maximum duration of 20 min. An additional volume of 300 mL has to be drunk in the 3 h after the meal. In both meals, at intervals of 30 min for a total of 3 h, a battery of Visual Analogue Scales (VAS) will be administered to assess possible differences in the satiating power of the two pizzas and their sensory characteristics, as described in the dedicated session.

Blood samples will be drawn from an indwelling antecubital venous cannula for the measurement of glucose, insulin and sodium concentration in the fasting state and every 30 min thereafter for 3 h after eating was begun and the Area Under the Curve will be calculated.

The volume of the 3 h urine collection will be measured, and the sodium and creatinine concentrations measured by ISE and by an enzymatic colorimetric method.

ELIGIBILITY:
Inclusion Criteria:

* 18 years,
* healthy volunteers

Exclusion Criteria:

* smoking,
* hypertension,
* diabetes,
* hyperlipidemia,
* eating disorders,
* use of medications affecting satiety and hunger sensations,
* past gastrointestinal surgery potentially affecting digestion and absorption processes,
* presence of chronic diseases
* strenuous physical activity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of sensory characteristics of the pizza | 20 minutes
  Administration of a Visual Analogue Scale (VAS) just after the meal for testing the following four sensory characteristics: chewness, flavour, saltiness, general pleasantness
Evaluation of the satiating power of the pizza | 3 hours
  Administration of a Visual Analogue Scale (VAS) for a 3 hours period for testing the followings: hunger, satiety, desire to eat more pizza, prospective to eat more

SECONDARY OUTCOMES:
Evaluation of the metabolic response of the study participants (glucose) | 3 hours
  Evaluation of changes in glucose parameters. Blood samples will be drawn from an indwelling antecubital venous cannula for the measurement of glucose concentration in the fasting state and every 30 min thereafter for 3 h after eating is begun. Serum glucose level will be measured by an enzymatic colorimetric method (Pentra 400, Horiba ABX, Rome, Italy), and tha area under the curve will be calculated.
Evaluation of the metabolic response of the study participants (insulin) | 3 hours
  Evaluation of changes in insulin parameters. Blood samples will be drawn from an indwelling antecubital venous cannula for the measurement of insulin concentration in the fasting state and every 30 min thereafter for 3 h after eating is begun, Serum insulin concentration will be measured by ELISA (DIA source, Dusseldorf, Germany) and the area under the curve will be calculated.
Evaluation of sodium metabolism | 3 hours
  Blood samples will be drawn from an indwelling antecubital venous cannula for the measurement of sodium concentration in the fasting state and every 30 min thereafter for 3 h after eating was begun. Plasma sodium concentration will be measured by an ion-selective electrode (ISE) method (Pentra 400, Horiba ABX, Rome, Italy) and the Area Under the Curve will be calculated.
Evaluation of the sodium excretion | 3 hours
  The volume of the 3 h urine collection will be measured, and the sodium and creatinine concentrations will be measured by ISE and by an enzymatic colorimetric method. Urinary sodium excretion will be calculated in grams.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Strazzullo, MD, Principal Investigator — Federico II University
Locations (1):
- Federico II University Hospital, Napoli, Italy